CLINICAL TRIAL: NCT04485247
Title: Is Transumbilical Laparoscopy-assisted Appendectomy in the Pediatric Acute Uncomplicated Appendicitis Superior to Conventional 3 Port Laparoscopic Appendectomy?
Brief Title: Transumbilical Laparoscopy-assisted Appendectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Myongji Hospital (Other)
Responsible Party: Principal Investigator, Kyung-Goo Lee, Assistant professor, Myongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Myongji Surgery
Record Dates: First submitted 2020-07-20; First posted 2020-07-24 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Appendicitis Acute
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (Active Comparator): conventional laparoscopic appendectomy with 3-ports
  Interventions: Procedure: 3-port laparoscopic appendectomy
- TULAA group (Experimental): An operator extracts and ligates appendix through umbilical port.
  Interventions: Procedure: Transumbilical Laparoscopic-Assisted Appendectomy

INTERVENTIONS:
Procedure: Transumbilical Laparoscopic-Assisted Appendectomy — appendectomy performed extracorporeally through umbilical port
  Arms: TULAA group
Procedure: 3-port laparoscopic appendectomy — appendectomy performed intracorporeally with 3-port
  Arms: Conventional group

SUMMARY:
transumbilical laparoscopic-assisted appendectomy (TULAA) was reported that the operation time was shorter and the postoperative frequency of complications was not high compared to conventional laparoscopic appendectomy (CLA) with three conventional ports in retrospective studies. The purpose of this study is to evaluate the outcomes of transumbilical laparoscopic-assisted appendectomy (TULAA) and to compare them to the outcomes of CLA.

DETAILED DESCRIPTION:
Single port appendectomy can be considered as the better option than conventional laparoscopic appendectomy (CLA) for pediatric patients with uncomplicated acute appendicitis in cosmetic aspect. However, this technique has not gained popularity because it has been regarded as a tricky and time-consuming procedure. Recently, the frequency of implementation of transumbilical laparoscopy-assisted appendectomy (TULAA) is increasing in pediatric patients with uncomplicated appendicitis. The reason that this operation is possible in children, is that the length between umbilicus and appendix is shorter than that of an adult, and the abdominal wall is flexible, so that the appendix can be extracted through umbilical incision. It was reported that the operation time was shorter and the postoperative frequency of complications was not high compared to the laparoscopic appendectomy with three conventional ports. The purpose of this study is to evaluate the outcomes of transumbilical laparoscopic-assisted appendectomy (TULAA) and to compare them to the outcomes of CLA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically diagnosed as acute appendicitis
* Age 18 or under
* Lab tests Hemoglobin ≥ 10g/dl White blood cell count ≥ 4,000/mm3 Platelet count ≥ 100,000/mm3 Creatinine ≤ 1.5 mg/dl Aspartate aminotransferase ≤ 100 IU/L Alanine aminotransferase ≤ 100 IU/L
* no significant dysfunction in the heart, lungs, kidneys.

Exclusion Criteria:

* Previous abdominal operation
* Generalized peritonitis
* Anticipated extended resection
* Periappendiceal abscess on preoperative exam

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Operation time | 1 day
  Time from skin incision to skin closure

SECONDARY OUTCOMES:
Postoperative complication rate | 1 month
  Rate of 30 day complication or in-hospital complication
postoperative hospital stay | 1 month
  postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Goo Lee, MD, Principal Investigator — Myongji Hospital
Locations (1):
- Myongji Hospital, Hanyang university college of medicine, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: all individual participant data that underlie results in a publication

REFERENCES:
- [Background] Sekioka A, Takahashi T, Yamoto M, Miyake H, Fukumoto K, Nakaya K, Nomura A, Yamada Y, Urushihara N. Outcomes of Transumbilical Laparoscopic-Assisted Appendectomy and Conventional Laparoscopic Appendectomy for Acute Pediatric Appendicitis in a Single Institution. J Laparoendosc Adv Surg Tech A. 2018 Dec;28(12):1548-1552. doi: 10.1089/lap.2018.0306. Epub 2018 Aug 8. PMID 30088968
- [Result] Dubbers M, Nikolaou E, Fuchs H, Fischer J, Alakus H, Leers J, Bruns C, Cernaianu G. Update on Transumbilical Single-Incision Laparoscopic Assisted Appendectomy (TULAA) - Which Children Benefit and What are the Complications? Klin Padiatr. 2018 Jul;230(4):194-199. doi: 10.1055/s-0044-101622. Epub 2018 Mar 15. PMID 29544230
- [Result] Shekherdimian S, DeUgarte D. Transumbilical laparoscopic-assisted appendectomy: an extracorporeal single-incision alternative to conventional laparoscopic techniques. Am Surg. 2011 May;77(5):557-60. doi: 10.1177/000313481107700513. PMID 21679587